CLINICAL TRIAL: NCT02797561
Title: A Multicenter, Prospective Cohort to Evaluate the Effect of FFR Guided Percutaneous Coronary Intervention in Coronary Tandem Lesions
Brief Title: Effect of FFR Guided Percutaneous Coronary Intervention in Coronary Tandem Lesions
Acronym: IRISFFRTandem
Status: Recruiting | Type: Observational
Sponsor: Seung-Jung Park (Other)
Collaborators: CardioVascular Research Foundation, Korea (Other)
Responsible Party: Sponsor-Investigator, Seung-Jung Park, professor of medicine, Asan Medical Center
Organization: Asan Medical Center (Other)
Other Study IDs: AMCCV2016-12
Record Dates: First submitted 2016-06-08; First posted 2016-06-13 (Estimated); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Percutaneous Transluminal Coronary Angioplasty
Keywords: Fractional flow reserve; Tandem; Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Tandem lesion evaluated by FFR
  Interventions: Other: 5 year Follow-up

INTERVENTIONS:
Other: 5 year Follow-up

SUMMARY:
The purpose of this study is to evaluate the effect of FFR (Fractional flow reserve) guided Percutaneous Coronary Intervention in coronary tandem lesions.

ELIGIBILITY:
Inclusion Criteria:

* Tandem lesion evaluated by FFR
* Written consent

Exclusion Criteria:

* TIMI flow < 3
* Grafted vessel
* Left ventricular ejection fraction < 30%
* Severe calcification and/or severe tortuosity
* Uncontrolled coronary spasm
* Life expectancy < 2 years
* Planned high risk surgery
* Pregnancy or breast-feeding

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with tandem lesion evaluated by FFR
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2016-07-25 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure | 2 years
  defined as composite event of cardiac death, non-fatal myocardial infarction, target vessel revascularization

SECONDARY OUTCOMES:
all cause death | 5 years
cardiac death | 5 years
myocardial infarction | 5 years
target vessel revascularization | 5 years
target lesion revascularization | 5 years
Cardiac rehospitalization | 5 years
Cardiac death and myocardial infarction | 5 years
death, myocardial lnfarction, revascularization | 5 years
  related with stented lesion
stroke | 5 years
stent thrombosis | 5 years
angina | 5 years
number of antianginal medications | 5 years
complications with FFR | 5 years
clinical predictors of events | 5 years
functional index | 5 years
  IMR(index of microcirculatory resistance), CFR(CFRthermo)

CONTACTS AND LOCATIONS:
Locations (14):
- South Korea (14):
  - Asan Medical Center, Seoul, Songpa-gu
  - Soon Chun Hyang University Hospital Bucheon, Bucheon-si
  - Gangwon National Univ. Hospital, Chuncheon
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - Inje University Ilsan Paik Hospital, Ilsan
  - Bundang CHA Hospital, Seongnam
  - Seoul National University Bundang hospital, Seongnam
  - Kangbuk Samsung Hospital, Seoul
  - Seoul National University hospital, Seoul
  - Wonju Severance Christian Hospital, Wŏnju
  - Pusan National University Yangsan Hospital, Yangsan

IPD SHARING:
Plan to Share IPD: Undecided